CLINICAL TRIAL: NCT06096506
Title: Nourishing the Community Through Culinary Medicine- Acres Homes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: National Cancer Institute (NCI) (NIH); M.D. Anderson Cancer Center (Other)
Responsible Party: Principal Investigator, Natalia Heredia, Assistant Professor, The University of Texas Health Science Center, Houston
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: HSC-SPH-23-0810; 1U54CA280804-01 (NIH)
Record Dates: First submitted 2023-10-17; First posted 2023-10-23 (Actual); Last update posted 2024-12-06 (Actual); Status verified 2024-12

CONDITIONS: Diabetes; Elevated Body Mass Index
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention clinics (Experimental): Participants will be recruited from those receiving care at University of Texas (UT) Physician Clinics serving the Acres Homes neighborhood in Houston
  Interventions: Behavioral: Virtual Culinary Medicine
- Control Clinics (No Intervention): Participants will be recruited from UT Physicians clinics outside of the Acres Homes service area

INTERVENTIONS:
Behavioral: Virtual Culinary Medicine — The virtual curriculum will include five 90-minute sessions (to be held weekly or bi-weekly). Participants will also be expected to shop for groceries ahead of the sessions to participate in the program. A gift card will be provided for groceries ($30 per class = $150 total).Asynchronous virtual educational content (cooking skills videos, animated nutrition education videos, and additional recipes) will be provided to engage and retain participants beyond initial sessions
  Arms: Intervention clinics

SUMMARY:
The purpose of this study is to to implement adapted virtual Culinary Medicine (CM) curriculum among target population, to assess if program participation improves participant dietary behaviors, nutrition knowledge, and cooking skills and behaviors above standard of care, to assess if program participation improves patient levels of HbA1c, Body Mass Index, Blood Pressure, HDL, LDL and Triglycerides above standard of care and to determine the feasibility and reproducibility of virtual synchronous CM classes.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care at UT Physicians clinics
* diagnosed with type 2 diabetes and elevated body mass index (>=25)
* HbA1c labs and clinic-assessed weight completed within the last 3 months;
* English speaking or Spanish speaking.
* Can obtain groceries before each class (intervention group only)

Exclusion Criteria:

* Patients without the technological support needed to participate (e.g., reliable internet and device - cell phone, tablet or laptop);
* Patients with an uncontrolled impairment that interferes with ability to participate.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-10-30 (Actual)

PRIMARY OUTCOMES:
Change in Hemoglobin A1c (HbA1c) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)

SECONDARY OUTCOMES:
Change in Body Mass Index | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in systolic Blood Pressure | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in diastolic Blood Pressure | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in High-density lipoprotein (HDL) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in low-density lipoprotein (LDL) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in Triglyceride | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
Change in perceived health as assessed by the Nourishing the Community Through Culinary Medicine survey (NCCM | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This is a 1 item questionnaire and is scored from 1(excellent) to 6(poor) for a maximum score of 6, a higher number indicating better health
Change in fruit and vegetable consumption as assessed by the Nourishing the Community Through Culinary Medicine survey (NCCM | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This is a 2 item questionnaire and is scored from 0(no servings per day ) to 5(4+ servings per day), maximum score of 10 a higher number indicating more consumption of fruit and vegetables
Change in whole grain consumption as assessed by the Nourishing the Community Through Culinary Medicine survey (NCCM | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This is a 1 item questionnaire and is scored from 0(no servings per day ) to 5(4+ servings per day), maximum score of 5 a higher number indicating more consumption of whole grains
Change in typical food consumption behaviors as assessed by the Nourishing the Community Through Culinary Medicine survey (NCCM | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This consists of 7 items that are scored from 1 [Not at all] to 5 [More than once a day] for a maximum score of 35, a higher number indicating better outcome.
Change in Perceived Barriers of Eating Fruits and Vegetables as assessed by the Nourishing the Community Through Culinary Medicine survey (NCCM | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This consists of 13 items that are scored from 0( strongly agree) to 4( strongly disagree) for a maximum score of 52, a higher number indicating better outcome
Change in Eating/cooking/using nutrition labels by the Nourishing the Community Through Culinary Medicine survey (NCCM) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This consists of 10 items that are scored from 1( never) to 5( always) for a maximum score of 50, a higher number indicating better outcome
Change in Barriers to Healthy Eating by the Nourishing the Community Through Culinary Medicine survey (NCCM) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This consists of 4 items that are scored from 1( strongly agree) to 5( strongly disagree) for a maximum score of 20, a higher number indicating better outcome
Change in Self-efficacy in cooking food and meal planning by the Nourishing the Community Through Culinary Medicine survey (NCCM) | baseline (within 90 days of starting the NCCM program), at program completion (within 90 days of NCCM program completion)
  This consists of 5 items that are scored from 0( not at all sure) to 4( extremely sure ) for a maximum score of 20, a higher number indicating more self efficacy
Change in Diabetes Management by the Nourishing the Community Through Culinary Medicine survey (NCCM) | Baseline, post intervention (upto 10 weeks after baseline)
  This consists of 18 items. The first 16 items that are scored from 1 [Does not apply to me] to 4 [Applies to me very much] and the remaining 2 items are dichotomous scored [Yes=1] to [No=0], for a maximum score of 68, with a higher number indicates a better diabetes self-management.

CONTACTS AND LOCATIONS:
Overall Officials: Natalia I Heredia, PhD., MPH, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No